CLINICAL TRIAL: NCT06133491
Title: A Multi-Center Unblinded Proof-of-Concept Study of DaxibotulinumtoxinA for Migraine Prevention in High-Frequency and Chronic Migraine: the Standard Paradigm
Brief Title: Open Label, 6-month Study for High Frequency and Chronic Migraine,
Status: Active, not recruiting | Type: Observational
Sponsor: Ki Health Partners. LLC (Industry)
Collaborators: The Los Angeles Headache Center (Unknown); Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REV-002 Standard Paradigm
Record Dates: First submitted 2023-11-03; First posted 2023-11-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Daxibotulinumtonix A — SQ injections of 10u per site will be given over standard landmarks (18 sites) to patients who consent and are found eligible.

SUMMARY:
This is a prospective, multi-center, unblinded study in patients with migraine (≥ 8 MMDs/month) requiring preventive treatment. Enrolled patients will receive DAX administered subcutaneously using an established, published, legacy injection paradigm (referred to herein as the "standard paradigm"). The safety and efficacy outcome measures will be assessed at selected dosing segments during the 24-week treatment phase.

DETAILED DESCRIPTION:
Patients enrolled who meet eligibility will receive a total of 310 units of DAXI Injections in divided doses over 31 landmarks (sites), including the face, head, neck and shoulders, as identified per the standard paradigm, at visit 2. Follow-up visits via combination of phone and in office will occur at V3, week 8, through V9, week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from the subject in accordance with requirements of the study site's IRB or ethics committee, prior to initiation of any protocol-specified procedures.
2. Subject must be able to read.
3. Male or female subjects, 18 to 75 years of age inclusive.
4. Subject has at least a 1-year history of migraine (with or without aura) consistent with a diagnosis according to ICHD, 3rd edition with the following:

   * Age of onset prior to 50 years of age
   * Migraine attacks lasting on average 4-72 hours untreated.
   * By subject report at least 8 migraine days of moderate or severe intensity per month over the previous 3 months (prior to screening)
   * Ability to distinguish migraine from non-migraine headache.
   * No more than 26 headache days of any type per month by subject report.
5. Patients with at least 8 qualified migraine days per month over the three months prior to Screening will be eligible for entry into this study (assessed by historical recall). A migraine attack must last at least 30 minutes. Any use of an acute migraine-specific medication will count as a migraine attack (day). The interval between two qualified migraine days should be at least 24 hours to be counted as distinct migraine attacks. A migraine attack that remits following treatment (or sleep) and recurs within 24 hours will be counted as one migraine attack.
6. Females should be either of non-childbearing potential by reason of surgery, radiation, menopause (one year post onset), or of childbearing potential and practicing a medically acceptable method of contraception (eg, abstinence, a barrier method plus spermicide, or IUD) for at least one month before study randomization and for two months after the end of the study. Pregnant and/or lactating females are excluded. Those women using hormonal contraceptives must also be using an additional approved method of contraception (eg, a barrier method plus spermicide, or IUD) starting with the Baseline Phase and continuing throughout the entire study period.
7. A sub-set of subjects (capped at 30% of total enrolled) on not more than 1 preventive migraine medication may remain on therapy if the dose has been stable for at least 3 months (12 weeks) prior to the observation period and is not expected to change.

   * Exceptions include onobotulinumtoxinA treatment (wash out = 3 months).
   * Patients who are able and willing to attend study visits, maintain a headache diary and otherwise comply with study related activities.
   * Patients may be naive to BoNT therapy (no minimum or cap) or have received BoNT therapy provided there is a 3-month washout period.
   * A minimum of 30% of eligible subjects will be Chronic Migraine, per ICHD-3 criteria.

Exclusion Criteria:

1. Migraine patients with ≥26 headache days of any kind per month by historical report over the 3 months prior to study.
2. Patients with cluster headaches and other trigeminal autonomic cephalalgias, and other primary headaches (except tension-type headache) and secondary headaches (defined according to the Headache Classification Committee of the IHS, 3rd Edition, 2018),
3. Patients with a history of being non-responsive to adequate trials of more than two classes of migraine preventive treatments (e.g., beta blockers, calcium channel blockers, tricyclics, divalproex, topiramate, small or large molecule CGRP antagonists or onobotulinumtoxinA).
4. Patients who use the following medications as described:

   * Use of triptans, ditans or ergot-containing medications for 10 days or greater per month on average,
   * Use of NSAIDs, acetaminophen or combination analgesics (such as acetaminophen-caffeine products) 15 days or greater per month on average,
   * Use of opioids and/or butalbital containing medications for 4 days or greater per month on average,
   * Use of any two or more of the above medications (excluding opioids/butalbital) for 15 days or greater per month on average.
5. Patients with clinically significant neurological illness, other than migraine, that, in the opinion of the Investigators, may have the potential of altering pain perception or reporting,
6. Known or suspected serious neuromuscular, respiratory or cardiovascular disorder (such as amyotrophic lateral sclerosis, myasthenia gravis, severe chronic obstructive pulmonary disorder, coronary artery disease) that in the opinion of the investigator would place the participant at increased risk of an adverse event.
7. Patients with a history of or currently having major psychiatric disorders including schizophrenia, active psychosis or bipolar disorder. Major depressive disorder and generalized anxiety disorder which, in the investigator's opinion are well-controlled, will be allowed.
8. Patients with clinically significant active hepatic disease, cardiovascular, metabolic, respiratory, renal, endocrinological (including poorly controlled diabetes mellitus), gastrointestinal diseases, and bacterial or viral infections within 30 days prior to Screening or during the Baseline Phase, that in the opinion of the investigator may interfere with subject's participation in the study or may present a risk of the subject not completing the study.
9. Patients with hematologic or solid malignancy diagnosis within 5 years prior to screening with the exception of basal cell carcinoma and squamous cell carcinoma if they have been cancer free prior to screening.
10. Body mass index of <18 or >35.
11. Patients who within the past 3 years have a history of or have been treated for alcohol or drug abuse.
12. Women who are unwilling or unable to use acceptable contraception during the study.
13. Women who are pregnant or breastfeeding.
14. Patients who have participated in a drug intervention study for any indication within 60 days (or 5 half-lives of the investigational drug, whichever is longer) or non-drug intervention study (such as electrical stimulation) within 30 days.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and Women 18-75 years old with migraines (≥ 8 MMDs/month) requiring preventive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in monthly migraine days over weeks 9-12 as determined by patients reported outcomes on the daily headache diary. | Over weeks 9-12 (4 week period)

SECONDARY OUTCOMES:
Change from baseline in monthly migraine days over weeks 5-8 | 4 weeks - Over weeks 5-8
  Time to wear-off that would qualify the patient for retreatment.
The percentage of patients with a ≥50% reduction from baseline in monthly migraine days over weeks 9-12. | 4 weeks - Over weeks 9-12
  Time to wear-off that would qualify the patient for retreatment.
The percentage of patients with a ≥75% and 100% reduction from baseline in monthly migraine days over weeks 9-12. | 4 weeks - over weeks 9-12
  Time to wear-off that would qualify the patient for retreatment.
Change from baseline in the mean monthly migraine headache days requiring acute medication use to treat a migraine or headache across weeks 9-12. | 4 weeks - over weeks 9-12
  Time to wear-off that would qualify the patient for retreatment.
Change from baseline in the MIDAS score at week 12. | Week 12
  Time to wear-off that would qualify the patient for retreatment.
Change from baseline in the PGIC at multiple time points during 6 month study | over duration of study (6 months)
  Time to wear-off that would qualify the patient for retreatment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Los Angeles Headache Center, Los Angeles, California
  - New England Institute for Clinical Research, Stamford, Connecticut

IPD SHARING:
Plan to Share IPD: Undecided